CLINICAL TRIAL: NCT04628624
Title: The Effect of Green Tea Supplementation Strategies on Fat Oxidation and Body Composition in Overweight Individuals
Brief Title: Green Tea Supplementation, Fat Oxidation and Body Composition in Overweight Individuals
Acronym: GreenTea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anglia Ruskin University (Other)
Responsible Party: Principal Investigator, Justin Roberts, Associate Professor, Anglia Ruskin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: FST/FREP/17/703
Record Dates: First submitted 2020-11-05; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Overweight and Obesity; Fat Burn
Keywords: Green Tea; Exercise Metabolism
MeSH Terms: conditions — Overweight; Obesity | interventions — Antioxidants

STUDY DESIGN:
Intervention Model Description: Participants randomly assigned to either placebo, green tea extract (GTE) or GTE with antioxidants in a parallel, double blind manner
Who Masked: Participant, Investigator
Masking Description: Nutritional supplements will be provided in a randomised, double-blinded manner. Both the participants and research testers will be masked from knowing the specifics of the supplement intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Placebo Comparator): Placebo - capsulated, colour matched potato starch (~450mg per capsule) - provided by Biocare Ltd., UK using standard 00 vegetable capsules (hydroxypropyl methylcellulose). Dosage: 2 divided doses (1 capsule mid morning, 1 capsule mid afternoon) - daily for 8 weeks.
  Interventions: Dietary Supplement: Placebo control
- Green tea 1 (Experimental): Capsulated decaffeinated green tea extract (dGTE) (standardised to 70% EGCG concentration, 571mg total per day, containing 400mg EGCG - provided by Biocare Ltd., UK using standard 00 vegetable capsules (hydroxypropyl methylcellulose). Dosage: 2 divided doses (1 capsule mid morning, 1 capsule mid afternoon) - daily for 8 weeks.
  Interventions: Dietary Supplement: GTE 1
- Green tea 2 (Experimental): Capsulated decaffeinated green tea extract (dGTE) (standardised to 70% EGCG concentration, 571mg total per day, containing 400mg EGCG + 150mg quercitin and 150mg alpha lipoic acid - provided by Biocare Ltd., UK using standard 00 vegetable capsules (hydroxypropyl methylcellulose). Dosage: 2 divided doses (1 capsule mid morning, 1 capsule mid afternoon) - daily for 8 weeks.
  Interventions: Dietary Supplement: GTE 2

INTERVENTIONS:
Dietary Supplement: Placebo control — 8 week supplementation period, with participants consuming 2 capsules per day containing potato starch
  Other Names: Placebo
  Arms: Placebo group
Dietary Supplement: GTE 1 — 8 week supplementation period, with participants consuming 2 capsules per day containing green tea extract (571mg/d)
  Other Names: Decaffeinated green tea extract
  Arms: Green tea 1
Dietary Supplement: GTE 2 — 8 week supplementation period, with participants consuming 2 capsules per day containing green tea extract with additional antioxidants (150mg of quercitin and 150mg of alpha lipoic acid)
  Other Names: Decaffeinated green tea extract and antioxidants
  Arms: Green tea 2

SUMMARY:
The purpose of this study is to investigate the effects of green tea extract (GTE) on fat oxidation, body composition and exercise performance in overweight individuals. The study will be conducted under laboratory conditions following an 8 week supplemental period. Participants will be required to attend the laboratory for a pre-screening/familiarisation trial followed by assessments at week 0 (baseline), week 2, 4 and 8. Across the intervention, participants will maintain habitual dietary intake and follow a prescribed exercise programme. Additionally participants will be randomised to either a placebo, green tea extract or GTE with antioxidant supplementation.

It is hypothesised that the addition of antioxidants with GTE will enhance fat oxidation in overweight individuals more than GTE or placebo. It is further hypothesised that such improvements in fat oxidation due to GTE will lead to improvements in both body composition variables and submaximal exercise performance (metabolic efficiency) in overweight, but otherwise healthy persons.

DETAILED DESCRIPTION:
The health benefits of polyphenols found in green tea (GT), the unfermented leaves of the tea plant, Camellia sinensis, are of current scientific interest. These health benefits, in part, relate to the bioactive catechin polyphenol content of GT, of which (-)-epigallocatechin-3-gallate (EGCG) can account for between 50-80% of the total catechin content. GT catechins have been proposed to influence metabolic and thermogenic activities in the short term, leading to enhanced fat oxidation capacity, although this has been disputed.

Research investigating GT extracts (GTE) and exercise have produced conflicting results. Modest EGCG dosage in the short term (270 mg·d-1 EGCG for 6 days, and 68 mg·d-1 EGCG for 3 weeks) did not alter metabolic or performance variables in healthy or endurance trained volunteers. However, the inclusion of 100.5 mg·d-1 EGCG over a 10 week training period enhanced whole-body metabolic efficiency elsewhere. One confounding factor though is the use of caffeinated GTE in these studies. When decaffeinated GTE (dGTE) has been employed, 366 mg EGCG was found to acutely increase fat oxidation by 17%. Indeed a recent publication from our research group investigating the short term use of dGTE demonstrated positive changes in fat oxidation in healthy volunteers. However, less is known as to whether dGTE (or indeed combinations of dGTE with antioxidant nutrients which may improve GTE bioavailability) could provide similar results in overweight or sedentary individuals embarking on an exercise programme.

The aim of this research proposal is therefore to assess the impact of two GTE strategies on fat oxidation, cardiometabolic health, visceral fat reduction, and exercise performance in a healthy, but overweight cohort undertaking a standardised exercise training programme.

Research Questions:

Q1: Does regular consumption of dGTE favourably enhance fat oxidation and/or improve variables associated with cardiometabolic health and body composition in comparison to a placebo supplement in healthy, but overweight individuals? Q2: Does a dGTE complex (including key antioxidant nutrients) enhance fat oxidation and/or improve variables associated with cardiometabolic health and body composition more so than dGTE or placebo supplementation in healthy, but overweight individuals?

This study will involve participants attending sessions at Compass House, ARU, undertaking the following:

* Baseline trial: all participants will attend a subject briefing, provide written, informed consent prior to participation. Following this, all participants will undertake a baseline test for maximal fat oxidation rates (FATmax) and oxygen uptake using a standardised incremental cycling exercise protocol and expired air analysis
* Intervention period: participants will be randomly assigned to either dGTE (400mg EGCG daily), dGTE with antioxidants (150mg quercetin, 150mg alpha-lipoic acid) or placebo for 8 weeks. During this period, participants will undertake regular aerobic exercise (3x/ week; 45mins; at ~ FATmax intensity)
* Experimental evaluation of progress will be assessed at weeks 0,2,4, and 8. During laboratory visits, participants will be required to have a single venepuncture blood sample, assessment of blood pressure/ body composition (skinfold, bioelectrical impedance, waist circumference), assessment of FATmax, and assessment of fat oxidation during steady state exercise at FATmax.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, UK based, above 18 years of age
2. Below 45 years of age (for men) and below 55 years of age (for women)
3. Baseline maximal oxygen uptake >25ml/kg/min and <45ml/kg/min representative of normal (but not high) fitness levels; and a body mass index (BMI) >25kg/m2 and <33kg/m2
4. All participants: No known history (including family history) of heart abnormalities, hypertension, coronary heart disease or diabetes (determined from pre-study health screen questionnaire)
5. All participants: No known history of liver related disorders (e.g. hepatitis, Wilsons disease, cirrhosis).
6. All participants: Not currently suffering from any musculo-skeletal injury, or any other reason that may prevent participation in cardiovascular exercise
7. All participants: Have not suffered from recent viral infections ie: influenza (defined within the prior 2 months)
8. All participants: Not suffering from any known blood related disorders, including blood coagulation abnormalities, or have any adverse reactions to blood taking
9. All participants: Not taking any prescribed or over-the-counter medication which may influence exercise training (with the exception of inhalers for exercise induced asthma or contraceptive pill)
10. All participants: Not consuming or prepared to refrain from consumption, any commercial supplementation which conflicts with the study parameters ie: creatine, other green tea or weight loss products.

Exclusion Criteria:

1. Anyone below the age of 18 years, or above 45 years (for men) and 55 years (for women) - based on exercise testing guidelines by the American College of Sports Medicine (ACSM).
2. Those who do not meet the criteria for baseline maximal oxygen uptake or BMI assessment
3. All participants: anyone with a known history (including family history) of heart abnormalities, hypertension, coronary heart disease or diabetes (determined from pre-study health screen questionnaire)
4. All participants: anyone with a known previous history of liver related disorders.
5. All participants: Anyone suffering from a current musculo-skeletal injury, or any other reason that may prevent participation in cardiovascular exercise
6. All participants: those suffering from recent viral infections ie: influenza (defined within the prior 2 months)
7. All participants: Those with known blood related disorders, including blood coagulation abnormalities, or have any adverse reactions to blood taking. This includes any participant who has or potentially has an infectious disease, inc. HIV, and all types of hepatitis.
8. All participants: Anyone taking any prescribed or over-the-counter medication which may influence exercise training (with the exception of inhalers for exercise induced asthma or contraceptive pill)
9. All participants: Anyone consuming or not prepared to refrain from consumption, any commercial supplementation which conflicts with the study parameters ie: creatine, other green tea or weight loss products.
10. FEMALE ONLY: Any participant who is, suspects they may be or becomes pregnant during the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Fat oxidation (max) | Change from Baseline maximal fat oxidation at 1 month
  Assessment of maximal fat oxidation rate (via expired air) during incremental exercise
Fat oxidation (max) | Change from Baseline maximal fat oxidation at 2 months
  Assessment of maximal fat oxidation rate (via expired air) during incremental exercise
Fat oxidation (min) | Change from Baseline minimum fat oxidation at 1 month
  Assessment of exercise intensity at which point fat oxidation is negligable
Fat oxidation (min) | Change from Baseline minimum fat oxidation at 2 months
  Assessment of exercise intensity at which point fat oxidation is negligable

SECONDARY OUTCOMES:
Height | Change from baseline height at 1 month
  Assessment of height (in metres)
Height | Change from baseline height at 2 months
  Assessment of height (in metres)
Weight | Change from baseline weight at 1 month
  Assessment of weight (in kilograms)
Weight | Change from baseline weight at 2 months
  Assessment of weight (in kilograms)
Bodyfat percentage | Change from baseline bodyfat percentage at 1 month
  Assessment of bodyfat (%)
Bodyfat percentage | Change from baseline bodyfat percentage at 2 months
  Assessment of bodyfat (%)
Waist to hip ratio | Change from baseline waist to hip ratio at 1 month
  Assessment of waist to hip ratio (cm)
Waist to hip ratio | Change from baseline waist to hip ratio at 2 months
  Assessment of waist to hip ratio (cm)
Body mass index | Change from baseline BMI at 1 month
  Assessment of body mass index or BMI (measured in kilograms per metre squared)
Body mass index | Change from baseline BMI at 2 months
  Assessment of body mass index or BMI (measured in kilograms per metre squared)
Central abdomen depth | Change from baseline central abdominal depth at 1 month
  Assessment of central abdomen depth (in cm)
Central abdomen depth | Change from baseline central abdominal depth at 2 months
  Assessment of central abdomen depth (in cm)
Blood cholesterol | Change from Baseline at 1 month
  Assessment of total cholesterol, triglycerides, HDL-c and LDL-c (all in mmol/L)
Blood cholesterol | Change from Baseline at 2 months
  Assessment of total cholesterol, triglycerides, HDL-c and LDL-c (all in mmol/L)
Blood glucose | Change from Baseline blood glucose at 1 month
  Assessment of blood glucose (in mmol/L)
Blood glucose | Change from Baseline blood glucose at 2 months
  Assessment of blood glucose (in mmol/L)
Blood insulin | Change from Baseline blood insulin at 1 month
  Assessment of blood glucose (in pmol/L)
Blood insulin | Change from Baseline blood insulin at 2 months
  Assessment of blood glucose (in pmol/L)
Blood leptin | Change from Baseline blood leptin at 1 month
  Assessment of blood leptin (in ng/ml)
Blood leptin | Change from Baseline blood leptin at 2 months
  Assessment of blood leptin (in ng/ml)
Blood adiponectin | Change from Baseline blood adiponectin at 1 month
  Assessment of blood adiponectin (in ug/ml)
Blood adiponectin | Change from Baseline blood adiponectin at 2 months
  Assessment of blood adiponectin (in ug/ml)
Blood fatty acids and glycerol | Change from Baseline at 1 month
  Assessment of blood free fatty acids and glycerol (both in umol/L)
Blood fatty acids and glycerol | Change from Baseline at 2 months
  Assessment of blood free fatty acids and glycerol (both in umol/L)
Blood liver enzymes | Change from baseline at 1 month
  Assessment of blood liver enzymes including alanine aminotransferase(ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) (all measured in U/L)
Blood liver enzymes | Change from baseline at 2 months
  Assessment of blood liver enzymes including alanine aminotransferase(ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) (all measured in U/L)
Blood bilirubin | Change from baseline bilirubin at 1 month
  Assessment of blood concentration of bilirubin (in umol/L)
Blood bilirubin | Change from baseline bilirubin at 2 months
  Assessment of blood concentration of bilirubin (in umol/L)
Respiratory measures (oxygen, carbon dioxide) during steady state exercise | Change from baseline at 1 month
  Assessment of expired oxygen and carbon dioxide (in litres per minute)
Respiratory measures (oxygen, carbon dioxide) during steady state exercise | Change from baseline at 2 months
  Assessment of mean expired oxygen and carbon dioxide (in litres per minute)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Roberts, PhD, Principal Investigator — Anglia Ruskin University
Locations (1):
- Anglia Ruskin University, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roberts JD, Roberts MG, Tarpey MD, Weekes JC, Thomas CH. The effect of a decaffeinated green tea extract formula on fat oxidation, body composition and exercise performance. J Int Soc Sports Nutr. 2015 Jan 21;12(1):1. doi: 10.1186/s12970-014-0062-7. eCollection 2015. PMID 25650043
- [Background] Hursel R, Viechtbauer W, Westerterp-Plantenga MS. The effects of green tea on weight loss and weight maintenance: a meta-analysis. Int J Obes (Lond). 2009 Sep;33(9):956-61. doi: 10.1038/ijo.2009.135. Epub 2009 Jul 14. PMID 19597519
- [Background] Hursel R, Westerterp-Plantenga MS. Thermogenic ingredients and body weight regulation. Int J Obes (Lond). 2010 Apr;34(4):659-69. doi: 10.1038/ijo.2009.299. Epub 2010 Feb 9. PMID 20142827
- [Background] Ichinose T, Nomura S, Someya Y, Akimoto S, Tachiyashiki K, Imaizumi K. Effect of endurance training supplemented with green tea extract on substrate metabolism during exercise in humans. Scand J Med Sci Sports. 2011 Aug;21(4):598-605. doi: 10.1111/j.1600-0838.2009.01077.x. Epub 2010 Mar 10. PMID 20459475
- [Background] Venables MC, Hulston CJ, Cox HR, Jeukendrup AE. Green tea extract ingestion, fat oxidation, and glucose tolerance in healthy humans. Am J Clin Nutr. 2008 Mar;87(3):778-84. doi: 10.1093/ajcn/87.3.778. PMID 18326618
- [Background] Dulloo AG, Duret C, Rohrer D, Girardier L, Mensi N, Fathi M, Chantre P, Vandermander J. Efficacy of a green tea extract rich in catechin polyphenols and caffeine in increasing 24-h energy expenditure and fat oxidation in humans. Am J Clin Nutr. 1999 Dec;70(6):1040-5. doi: 10.1093/ajcn/70.6.1040. PMID 10584049
- [Background] Ryu OH, Lee J, Lee KW, Kim HY, Seo JA, Kim SG, Kim NH, Baik SH, Choi DS, Choi KM. Effects of green tea consumption on inflammation, insulin resistance and pulse wave velocity in type 2 diabetes patients. Diabetes Res Clin Pract. 2006 Mar;71(3):356-8. doi: 10.1016/j.diabres.2005.08.001. Epub 2005 Sep 19. PMID 16169629
- [Background] Maki KC, Reeves MS, Farmer M, Yasunaga K, Matsuo N, Katsuragi Y, Komikado M, Tokimitsu I, Wilder D, Jones F, Blumberg JB, Cartwright Y. Green tea catechin consumption enhances exercise-induced abdominal fat loss in overweight and obese adults. J Nutr. 2009 Feb;139(2):264-70. doi: 10.3945/jn.108.098293. Epub 2008 Dec 11. PMID 19074207
- [Background] Feng WY. Metabolism of green tea catechins: an overview. Curr Drug Metab. 2006 Oct;7(7):755-809. doi: 10.2174/138920006778520552. PMID 17073579
- [Background] Hodgson AB, Randell RK, Jeukendrup AE. The effect of green tea extract on fat oxidation at rest and during exercise: evidence of efficacy and proposed mechanisms. Adv Nutr. 2013 Mar 1;4(2):129-40. doi: 10.3945/an.112.003269. PMID 23493529
- [Background] Dean S, Braakhuis A, Paton C. The effects of EGCG on fat oxidation and endurance performance in male cyclists. Int J Sport Nutr Exerc Metab. 2009 Dec;19(6):624-44. doi: 10.1123/ijsnem.19.6.624. PMID 20175431
- [Background] Eichenberger P, Colombani PC, Mettler S. Effects of 3-week consumption of green tea extracts on whole-body metabolism during cycling exercise in endurance-trained men. Int J Vitam Nutr Res. 2009 Jan;79(1):24-33. doi: 10.1024/0300-9831.79.1.24. PMID 19839000
- [Background] Achten J, Jeukendrup AE. Maximal fat oxidation during exercise in trained men. Int J Sports Med. 2003 Nov;24(8):603-8. doi: 10.1055/s-2003-43265. PMID 14598198